CLINICAL TRIAL: NCT05000762
Title: Zinc Supplementation Improves Cardiovascular Morbidity in Patients With Diabetes Mellitus
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor no longer has support available.
Sponsor: Wayne State University (Other)
Collaborators: QPathology (Unknown)
Responsible Party: Principal Investigator, Warren Lockette, M.D., Professor of Medicine and Endocrinology, Wayne State University
Other Study IDs: IRB-20-10-2833
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
Keywords: Zinc dietary supplement; diabetes mellitus; cardiovascular reactivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus | interventions — Zinc

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diabetes mellitus: Patients with type 2 diabetes mellitus
  Interventions: Dietary Supplement: Zinc

INTERVENTIONS:
Dietary Supplement: Zinc — Zinc gluconate 30 mg/day orally

SUMMARY:
Oral zinc supplementation in patients with diabetes mellitus can improve glycemic control. However, there is reluctance to recommend zinc supplements to these patients because there is no evidence that the zinc-dependent improvement in glycemic control offers protections from the cardiovascular morbidities associated with diabetes mellitus, especially myocardial infarction and thrombotic stroke. The investigators are conducting a randomized, double blind, cross over study to test the hypothesis that oral zinc supplementation will block the enhanced cardiovascular, cerebrovascular, and platelet reactivity that lead to myocardial infarction and stroke in research participants with diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus induces adverse changes in the systemic blood vessels, the cerebral vasculature, and platelets that can culminate in myocardial infarction and thrombotic stroke. Also, when compared to patients whose diabetes mellitus is well controlled, poor glucose maintenance in men and women with diabetes mellitus undeniably confers a much greater risk of myocardial infarction and stroke. For these reasons, it is important to maintain euglycemia in patients with diabetes mellitus. Several studies have shown supplemention with oral zinc improves glycemic control in patients with diabetes mellitus. Zinc supplementation has been associated with an absolute fall in glycosylated hemoglobin (HgbA1c), a measurement of metabolic control, by 0.5 percentage points. It is unknown whether this dietary supplement improves the exaggerated systemic and cerebrovascular and platelet responsiveness that are responsible for the increased prevalence of myocardial infarction and stroke in patients with diabetes mellitus. The investigators postulate that zinc dietary supplementation, when compared to placebo, will significantly reduce the increased cardiovascular reactivity and thrombogenesis associated with myocardial infarction or stroke in men and women with diabetes mellitus. The investigators will conduct a randomized, double-blinded, cross over study in volunteers with diabetes mellitus in which the participants receive either four months of placebo or oral zinc gluconate (30 mg zinc gluconate). Subjects will have validated, non-invasive, non-pharmacologic assessments of both their systemic and cerebrovascular reactivity and platelet responsiveness. The investigators anticipate that zinc supplementation will enhance flow mediated endothelium-dependent vasodilation in the peripheral vasculature in patients with diabetes mellitus, and also, reduces cardiovascular responses to stress. It is expected that zinc supplementation will blunt the magnitude of blood pressure increases induced by exercise in the research subjects. Also, the investigators expect to show that zinc supplementation, when compared to placebo, reduces pulse wave velocity, a measure of vascular stiffness, in the research subjects with diabetes mellitus. The investigators will show that zinc supplementation, when compared to placebo, improves cerebral blood flow in patients with diabetes mellitus. The investigators will assess cerebrovascular reactivity by measuring the sensitivity of intracerebral blood vessels to increasing concentrations of pCO2, a maneuver which selectively relaxes the cerebral vasculature and increases cerebral blood flow. Finally, the investigators anticipate that zinc supplementation will reduce platelet aggregation.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with stable type 2 diabetes mellitus or pre-diabetes (HgbA1c between 6% - 9%) and who are otherwise healthy

Exclusion Criteria:

* Pregnant women
* Anyone unable to understand or give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women between the ages of 18 - 75 years who have stable type 2 diabetes or pre-diabetes reflected by a glycosylated heoglobin A1C between 6% - 9%. On no prescription medications other than for diabetes mellitus or nutritional supplements containing zinc
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | 4 months
  Measure changes non-invasively wtihcarotid-femoral pulse wave velocity
Cerebrovascular reactivity | 4 months
  Measure vasodilation in response to increasing pCO2
Blood pressure response to exercise | 4 months
  Assess blood pressure response to hand grip exercise
Platelet aggregation | 4 months
  Measure catecholamine-induced platelet aggregation ex vivo

CONTACTS AND LOCATIONS:
Overall Officials: Warren Lockette, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University School of Medicine, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Only anonymous, aggregate data will be shared, and only upon request.

REFERENCES:
- [Background] Jayawardena R, Ranasinghe P, Galappatthy P, Malkanthi R, Constantine G, Katulanda P. Effects of zinc supplementation on diabetes mellitus: a systematic review and meta-analysis. Diabetol Metab Syndr. 2012 Apr 19;4(1):13. doi: 10.1186/1758-5996-4-13. PMID 22515411